CLINICAL TRIAL: NCT05552560
Title: Access to Sperm Donation for Female Couples and Unmarried Women: First Descriptive Data at the Toulouse University Hospital. PLEIAD
Brief Title: Access to Sperm Donation for Female Couples and Unmarried Women
Acronym: PLEIAD
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0271
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Heterosexual couples, women or single women who have requested sperm donation: Heterosexual couples, female couples or single women who have requested a sperm donation in the center of the Toulouse University Hospital will be offered the study.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A questionnaire is offered to patients who meet the eligibility criteria and who have given their non-objection before the first consultation with the centre's psychologist.
  This questionnaire includes questions on the socio-demographic characteristics, the motivations, as well as the procreative history of the patients.

SUMMARY:
The Bioethics Law of August 2, 2021 now authorizes, in addition to heterosexual couples, access to sperm donation for female couples and unmarried women.

According to the Ministry of Health, since the opening of sperm donation to these new populations, requests at the national level (7000 during the first 6 months) have greatly exceeded the predicted figures (3000 per year). Welcoming this new patient population requires us, health professionals, to know it well. Indeed, to date, there is no reliable assessment in France of the life course, particularly reproductive, nor of the socio-demographic characteristics, nor of the psychological well-being of these patients.

This study via a pseudonymised questionnaire aims to fill this lack of information in order to help professionals build relevant care pathways.

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual couples, OR couples of women OR single women who have requested a sperm donation at the Center for Reproductive Medicine at the Toulouse University Hospital
* Patients who have given their consent (oral or written) after clear and fair information

Exclusion Criteria:

* First consultation with the centre's psychologist already carried out.
* Not fluent in French
* Protected adults (safeguard of justice, guardianship, curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heterosexual couples, women or single women who have requested sperm donation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Socio-demographic characteristics | Day 1
  Survey of socio-demographic characteristics of all persons eligible for sperm donation

CONTACTS AND LOCATIONS:
Overall Officials: Roger LEANDRI, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No